CLINICAL TRIAL: NCT02265029
Title: Evaluation of Spa Therapy in the Treatment of Fibromyalgia : a Randomized, Controlled, Open Multicenter Study
Brief Title: Evaluation of Spa Therapy in the Treatment of Fibromyalgia
Acronym: THERMALGI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association Francaise pour la Recherche Thermale (Other)
Collaborators: Floralis (Industry); University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DCIC/13/68
Record Dates: First submitted 2014-10-09; First posted 2014-10-15 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Fibromyalgia; Rheumatism, Muscular
Keywords: fibromyalgia; rheumatism; fatigue syndrom; pain; spa treatment in rheumatology
MeSH Terms: conditions — Fibromyalgia; Rheumatic Diseases; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate spa treatment (Active Comparator): Spa treatment during 18 days soon after randomization : the most adapted to the concerned pathology and common to all of spa resorts (whirpool bath with automatic air and water massage cycles, massaging shower,...)
  Interventions: Other: Immediate spa treatment
- Late SPA treatment (Sham Comparator): Spa treatment during 18 days soon after 6 months visit : the most adapted to the concerned pathology and common to all of spa resorts (whirpool bath with automatic air and water massage cycles, massaging shower,...)
  Interventions: Other: Late spa treatment

INTERVENTIONS:
Other: Immediate spa treatment — spa treatment in rheumatology with sedative and antalgique techniques and mobilizing techniques (rehabilitation in pool)
  Other Names: Spa treatment soon after randomisation
  Arms: Immediate spa treatment
Other: Late spa treatment — spa treatment in rheumatology with sedative and antalgique techniques and mobilizing techniques (rehabilitation in pool)
  Other Names: Spa treatment after 6 months visit in the study
  Arms: Late SPA treatment

SUMMARY:
Fibromyalgia is a common health problem that causes widespread pain and tenderness (sensitive to touch). The pain and tenderness tend to come and go, and move about the body. There is no cure for fibromyalgia. Complementary and alternative therapy such as acupuncture, chiropractic and massage therapy, can be useful to manage fibromyalgia symptoms. Many of these treatments have not been well tested in patients with fibromyalgia. Fibromyalgia affect 3 to 4% of the general population and 14 % of patients with rheumatologic disease. Fibromyalgia is most common in women 90 % in many studies. It most often starts in middle adulthood. A chronic evolution occured for Fibromyalgic patients with a major alteration of quality of life.

Thermalgi is a randomized, multicentre, open label trial wich aims to evaluate the effects of spa therapy in rheumatologia on evolution of disability in daily life of patients with fibromyalgia.

DETAILED DESCRIPTION:
THERMALGI is a controlled, randomized, multicentre, open label trial wich aims to evaluate the effects of spa therapy in rheumatologia on evolution of disability in daily life of patients with fibromyalgia.

Patients with fibromyalgia (American College of Rheumatology Criteria) and a FIQ score (Fibromyalgia Impact Questionnaire) > 39 will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* both sexes, more than 18 years old patients
* available for a spa treatment in rheumatology during 18 days (immediate or late spa) and a follow-up period of 12 months
* with fibromyalgia ( ACR criteria 2010) for at least 1 year and with a stable treatment for at least 3 months
* with a FIQ score > or = 39 (fibromyalgia moderate to severe)
* voluntary to participate to the study, informed consent form signed after appropriate information
* affiliation to the social security system or equivalent

Exclusion Criteria:

* contra-indication of spa treatment (cancer in progress, psychiatrics disorders, immunodeficiency)
* no previous spa treatment in rheumatology within 1 year prior to inclusion
* substantial variation of the therapeutic coverage in the previous 3 months the inclusion (change of medicinal class, starting up of a réentrainement in the effort or a cognitivio-behavioral technique)
* subject with an other chronic severe disease (severe asthma, severe cardiac insuffisiancy, respiratory, renal or liver failures, evolutive rheumatic disease, inflammatory colitis...)
* subject participating to an other clinical study inerventionnal
* pregnancy, parturient or breast feeding
* no psychiatric illness or social situation that would preclude study compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Handicap in everyday life | 6 months
  Decrease of 14% (success rate) of FIQ questionnaire at 6 months compare to baseline

SECONDARY OUTCOMES:
Quality of life | at baseline, 3, 6, 9 and 12 months
  1. Comparison of the FIQ questionnaire mean between baseline, 3 and 6 months. Quantitative evaluation of the primary outcome.
  2. EUROQUOL (EQ5D) score evolution between baseline, 6 and 12 months.
  3. Evolution of PGA (autoevaluation) (Patient Global Assessment) and IGA (hetero evaluation) (Investigator's Global Assessment) scores between baseline, 3, 6, 9 and 12 months.
Pain evolution | at baseline, 3, 6, 9 and 12 months
  Monthly evolution of VAS (Visual Analogic Scale) pain and PCS questionnaire (Pain Catastrophizing Scale) between baseline, 3, 6, 9 and 12 months
Sleep quality | at baseline, 3, 6, 9 and 12 months
  Evolution of PSQI questionnaire (Pittsburg Sleep Quality Index) and Epworth Scale (ESS) (Epworth Sleepiness Scale) between baseline, 3, 6, 9 and 12 months
Fatigue | at baseline, 3, 6, 9 and 12 months
  Evolution of Pichot questionnaire between baseline, 3, 6, 9 and 12 months
Depression | at baseline, 3, 6, 9 and 12 months
  Evolution of HADS (Hospital Anxiety Depression Scale) and Coping-Etat questionnaires between baseline, 3, 6, 9 and 12 months
Ability to cope | at baseline, 6 and 12 months
  Evolution of Coping-Etat questionnaire between baseline, 6 and 12 months
Physical activity | at baseline, 3, 6, 9 and 12 months
  1. Evolution of Baecke score between baseline, 3, 6, 9 and 12 months
  2. evolution of BMI (Bone Mass Index) between baseline, 3, 6, 9 and 12 months
Medico economic impact | at baseline, 3, 6, 9 and 12 months
  Drugs consumption, medical and paramedical consultations, hospitalisations, professional absenteeism, complementary medicines resort.
Objective physical activity | at baseline, 3, and 6 months
  Record of day activity during one week with actigraphy at baseline, 3 and 6 months
Objective sleep quality | at baseline, 3, and 6 months
  Record of night activity and cardiac variability at baseline, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Caroline MAINDET DOMINICI, MD, Principal Investigator — Hospital University Grenoble
Locations (5):
- France (5):
  - station thermale AIX LES BAINS, Aix-les-Bains
  - station thermale ALLEVARD LES BAINS, Allevard
  - station thermale BOURBON LANCY, Bourbon-Lancy
  - station thermale LAMALOU LES BAINS, Lamalou-les-Bains
  - Station thermale URIAGE LES BAINS, Uriage-les-Bains

REFERENCES:
- [Background] Adler GK, Kinsley BT, Hurwitz S, Mossey CJ, Goldenberg DL. Reduced hypothalamic-pituitary and sympathoadrenal responses to hypoglycemia in women with fibromyalgia syndrome. Am J Med. 1999 May;106(5):534-43. doi: 10.1016/s0002-9343(99)00074-1. PMID 10335725
- [Background] Altan L, Bingol U, Aykac M, Koc Z, Yurtkuran M. Investigation of the effects of pool-based exercise on fibromyalgia syndrome. Rheumatol Int. 2004 Sep;24(5):272-7. doi: 10.1007/s00296-003-0371-7. Epub 2003 Sep 24. PMID 14508601
- [Background] Arnold LM, Clauw DJ, Wohlreich MM, Wang F, Ahl J, Gaynor PJ, Chappell AS. Efficacy of duloxetine in patients with fibromyalgia: pooled analysis of 4 placebo-controlled clinical trials. Prim Care Companion J Clin Psychiatry. 2009;11(5):237-44. doi: 10.4088/PCC.08m00680. PMID 19956462
- [Background] Baranowsky J, Klose P, Musial F, Hauser W, Dobos G, Langhorst J. Qualitative systemic review of randomized controlled trials on complementary and alternative medicine treatments in fibromyalgia. Rheumatol Int. 2009 Nov;30(1):1-21. doi: 10.1007/s00296-009-0977-5. Epub 2009 Aug 12. PMID 19672601
- [Background] Bellometti S, Galzigna L. Function of the hypothalamic adrenal axis in patients with fibromyalgia syndrome undergoing mud-pack treatment. Int J Clin Pharmacol Res. 1999;19(1):27-33. PMID 10450540
- [Background] Bennett RM, Bushmakin AG, Cappelleri JC, Zlateva G, Sadosky AB. Minimal clinically important difference in the fibromyalgia impact questionnaire. J Rheumatol. 2009 Jun;36(6):1304-11. doi: 10.3899/jrheum.081090. Epub 2009 Apr 15. PMID 19369473
- [Background] Bennett RM, Kamin M, Karim R, Rosenthal N. Tramadol and acetaminophen combination tablets in the treatment of fibromyalgia pain: a double-blind, randomized, placebo-controlled study. Am J Med. 2003 May;114(7):537-45. doi: 10.1016/s0002-9343(03)00116-5. PMID 12753877
- [Background] Biasi G, Manca S, Manganelli S, Marcolongo R. Tramadol in the fibromyalgia syndrome: a controlled clinical trial versus placebo. Int J Clin Pharmacol Res. 1998;18(1):13-9. PMID 9604730
- [Background] Bircan C, Karasel SA, Akgun B, El O, Alper S. Effects of muscle strengthening versus aerobic exercise program in fibromyalgia. Rheumatol Int. 2008 Apr;28(6):527-32. doi: 10.1007/s00296-007-0484-5. Epub 2007 Nov 3. PMID 17982749
- [Background] Branco JC, Bannwarth B, Failde I, Abello Carbonell J, Blotman F, Spaeth M, Saraiva F, Nacci F, Thomas E, Caubere JP, Le Lay K, Taieb C, Matucci-Cerinic M. Prevalence of fibromyalgia: a survey in five European countries. Semin Arthritis Rheum. 2010 Jun;39(6):448-53. doi: 10.1016/j.semarthrit.2008.12.003. Epub 2009 Feb 27. PMID 19250656
- [Background] Burckhardt CS, Mannerkorpi K, Hedenberg L, Bjelle A. A randomized, controlled clinical trial of education and physical training for women with fibromyalgia. J Rheumatol. 1994 Apr;21(4):714-20. PMID 8035399
- [Background] Burckhardt CS. Multidisciplinary approaches for management of fibromyalgia. Curr Pharm Des. 2006;12(1):59-66. PMID 16454725
- [Background] Busch AJ, Schachter CL, Overend TJ, Peloso PM, Barber KA. Exercise for fibromyalgia: a systematic review. J Rheumatol. 2008 Jun;35(6):1130-44. Epub 2008 May 1. PMID 18464301
- [Background] Busch AJ, Barber KA, Overend TJ, Peloso PM, Schachter CL. Exercise for treating fibromyalgia syndrome. Cochrane Database Syst Rev. 2007 Oct 17;2007(4):CD003786. doi: 10.1002/14651858.CD003786.pub2. PMID 17943797
- [Background] Buskila D, Neumann L, Vaisberg G, Alkalay D, Wolfe F. Increased rates of fibromyalgia following cervical spine injury. A controlled study of 161 cases of traumatic injury. Arthritis Rheum. 1997 Mar;40(3):446-52. doi: 10.1002/art.1780400310. PMID 9082932
- [Background] Carville SF, Arendt-Nielsen L, Bliddal H, Blotman F, Branco JC, Buskila D, Da Silva JA, Danneskiold-Samsoe B, Dincer F, Henriksson C, Henriksson KG, Kosek E, Longley K, McCarthy GM, Perrot S, Puszczewicz M, Sarzi-Puttini P, Silman A, Spath M, Choy EH; EULAR. EULAR evidence-based recommendations for the management of fibromyalgia syndrome. Ann Rheum Dis. 2008 Apr;67(4):536-41. doi: 10.1136/ard.2007.071522. Epub 2007 Jul 20. PMID 17644548
- [Background] Cedraschi C, Desmeules J, Rapiti E, Baumgartner E, Cohen P, Finckh A, Allaz AF, Vischer TL. Fibromyalgia: a randomised, controlled trial of a treatment programme based on self management. Ann Rheum Dis. 2004 Mar;63(3):290-6. doi: 10.1136/ard.2002.004945. PMID 14962965
- [Background] Crofford LJ, Rowbotham MC, Mease PJ, Russell IJ, Dworkin RH, Corbin AE, Young JP Jr, LaMoreaux LK, Martin SA, Sharma U; Pregabalin 1008-105 Study Group. Pregabalin for the treatment of fibromyalgia syndrome: results of a randomized, double-blind, placebo-controlled trial. Arthritis Rheum. 2005 Apr;52(4):1264-73. doi: 10.1002/art.20983. PMID 15818684
- [Background] Dauvilliers Y, Touchon J. [Sleep in fibromyalgia: review of clinical and polysomnographic data]. Neurophysiol Clin. 2001 Feb;31(1):18-33. doi: 10.1016/s0987-7053(00)00240-9. French. PMID 11281066
- [Background] Evcik D, Kizilay B, Gokcen E. The effects of balneotherapy on fibromyalgia patients. Rheumatol Int. 2002 Jun;22(2):56-9. doi: 10.1007/s00296-002-0189-8. Epub 2002 Mar 29. PMID 12070676
- [Background] Donmez A, Karagulle MZ, Tercan N, Dinler M, Issever H, Karagulle M, Turan M. SPA therapy in fibromyalgia: a randomised controlled clinic study. Rheumatol Int. 2005 Dec;26(2):168-72. doi: 10.1007/s00296-005-0623-9. Epub 2005 Jun 17. PMID 15965635
- [Background] Fioravanti A, Perpignano G, Tirri G, Cardinale G, Gianniti C, Lanza CE, Loi A, Tirri E, Sfriso P, Cozzi F. Effects of mud-bath treatment on fibromyalgia patients: a randomized clinical trial. Rheumatol Int. 2007 Oct;27(12):1157-61. doi: 10.1007/s00296-007-0358-x. Epub 2007 May 23. PMID 17520260
- [Background] Forestier R, Desfour H, Tessier JM, Francon A, Foote AM, Genty C, Rolland C, Roques CF, Bosson JL. Spa therapy in the treatment of knee osteoarthritis: a large randomised multicentre trial. Ann Rheum Dis. 2010 Apr;69(4):660-5. doi: 10.1136/ard.2009.113209. Epub 2009 Sep 3. PMID 19734131
- [Background] Furlan R, Colombo S, Perego F, Atzeni F, Diana A, Barbic F, Porta A, Pace F, Malliani A, Sarzi-Puttini P. Abnormalities of cardiovascular neural control and reduced orthostatic tolerance in patients with primary fibromyalgia. J Rheumatol. 2005 Sep;32(9):1787-93. PMID 16142879
- [Background] Giske L, Vollestad NK, Mengshoel AM, Jensen J, Knardahl S, Roe C. Attenuated adrenergic responses to exercise in women with fibromyalgia--a controlled study. Eur J Pain. 2008 Apr;12(3):351-60. doi: 10.1016/j.ejpain.2007.07.007. Epub 2007 Sep 10. PMID 17827042
- [Background] Guetin S, Ginies P, Siou DK, Picot MC, Pommie C, Guldner E, Gosp AM, Ostyn K, Coudeyre E, Touchon J. The effects of music intervention in the management of chronic pain: a single-blind, randomized, controlled trial. Clin J Pain. 2012 May;28(4):329-37. doi: 10.1097/AJP.0b013e31822be973. PMID 22001666
- [Background] Hassett AL, Radvanski DC, Vaschillo EG, Vaschillo B, Sigal LH, Karavidas MK, Buyske S, Lehrer PM. A pilot study of the efficacy of heart rate variability (HRV) biofeedback in patients with fibromyalgia. Appl Psychophysiol Biofeedback. 2007 Mar;32(1):1-10. doi: 10.1007/s10484-006-9028-0. Epub 2007 Jan 12. PMID 17219062
- [Background] Jentoft ES, Kvalvik AG, Mengshoel AM. Effects of pool-based and land-based aerobic exercise on women with fibromyalgia/chronic widespread muscle pain. Arthritis Rheum. 2001 Feb;45(1):42-7. doi: 10.1002/1529-0131(200102)45:13.0.CO;2-A. PMID 11308060
- [Background] Kazlauskaite R, Evans AT, Villabona CV, Abdu TA, Ambrosi B, Atkinson AB, Choi CH, Clayton RN, Courtney CH, Gonc EN, Maghnie M, Rose SR, Soule SG, Tordjman K; Consortium for Evaluation of Corticotropin Test in Hypothalamic-Pituitary Adrenal Insufficiency. Corticotropin tests for hypothalamic-pituitary- adrenal insufficiency: a metaanalysis. J Clin Endocrinol Metab. 2008 Nov;93(11):4245-53. doi: 10.1210/jc.2008-0710. Epub 2008 Aug 12. PMID 18697868
- [Background] Kirschbaum C, Hellhammer DH. Salivary cortisol in psychoneuroendocrine research: recent developments and applications. Psychoneuroendocrinology. 1994;19(4):313-33. doi: 10.1016/0306-4530(94)90013-2. PMID 8047637
- [Background] Ledingham J, Doherty S, Doherty M. Primary fibromyalgia syndrome--an outcome study. Br J Rheumatol. 1993 Feb;32(2):139-42. doi: 10.1093/rheumatology/32.2.139. PMID 8428227
- [Background] Lerma C, Martinez A, Ruiz N, Vargas A, Infante O, Martinez-Lavin M. Nocturnal heart rate variability parameters as potential fibromyalgia biomarker: correlation with symptoms severity. Arthritis Res Ther. 2011;13(6):R185. doi: 10.1186/ar3513. Epub 2011 Nov 16. PMID 22087605
- [Background] McCain GA, Bell DA, Mai FM, Halliday PD. A controlled study of the effects of a supervised cardiovascular fitness training program on the manifestations of primary fibromyalgia. Arthritis Rheum. 1988 Sep;31(9):1135-41. doi: 10.1002/art.1780310908. PMID 3048273
- [Background] McCracken LM, MacKichan F, Eccleston C. Contextual cognitive-behavioral therapy for severely disabled chronic pain sufferers: effectiveness and clinically significant change. Eur J Pain. 2007 Apr;11(3):314-22. doi: 10.1016/j.ejpain.2006.05.004. Epub 2006 Jun 9. PMID 16762571
- [Background] McVeigh JG, McGaughey H, Hall M, Kane P. The effectiveness of hydrotherapy in the management of fibromyalgia syndrome: a systematic review. Rheumatol Int. 2008 Dec;29(2):119-30. doi: 10.1007/s00296-008-0674-9. Epub 2008 Aug 27. PMID 18751709
- [Background] Moldofsky H, Inhaber NH, Guinta DR, Alvarez-Horine SB. Effects of sodium oxybate on sleep physiology and sleep/wake-related symptoms in patients with fibromyalgia syndrome: a double-blind, randomized, placebo-controlled study. J Rheumatol. 2010 Oct;37(10):2156-66. doi: 10.3899/jrheum.091041. Epub 2010 Aug 3. PMID 20682669
- [Background] Moldofsky H, Lue FA, Mously C, Roth-Schechter B, Reynolds WJ. The effect of zolpidem in patients with fibromyalgia: a dose ranging, double blind, placebo controlled, modified crossover study. J Rheumatol. 1996 Mar;23(3):529-33. PMID 8832997
- [Background] Morley S, Williams ACC. RCTs of psychological treatments for chronic pain: progress and challenges. Pain. 2006 Apr;121(3):171-172. doi: 10.1016/j.pain.2006.01.017. Epub 2006 Mar 2. No abstract available. PMID 16513271
- [Background] Mostoufi SM, Afari N, Ahumada SM, Reis V, Wetherell JL. Health and distress predictors of heart rate variability in fibromyalgia and other forms of chronic pain. J Psychosom Res. 2012 Jan;72(1):39-44. doi: 10.1016/j.jpsychores.2011.05.007. Epub 2011 Jun 30. PMID 22200521
- [Background] Nater UM, Rohleder N. Salivary alpha-amylase as a non-invasive biomarker for the sympathetic nervous system: current state of research. Psychoneuroendocrinology. 2009 May;34(4):486-96. doi: 10.1016/j.psyneuen.2009.01.014. Epub 2009 Feb 26. PMID 19249160
- [Background] Onieva-Zafra MD, Castro-Sanchez AM, Mataran-Penarrocha GA, Moreno-Lorenzo C. Effect of music as nursing intervention for people diagnosed with fibromyalgia. Pain Manag Nurs. 2013 Jun;14(2):e39-46. doi: 10.1016/j.pmn.2010.09.004. Epub 2010 Nov 26. PMID 23108015
- [Background] Ozkurt S, Donmez A, Zeki Karagulle M, Uzunoglu E, Turan M, Erdogan N. Balneotherapy in fibromyalgia: a single blind randomized controlled clinical study. Rheumatol Int. 2012 Jul;32(7):1949-54. doi: 10.1007/s00296-011-1888-9. Epub 2011 Apr 2. PMID 21461716
- [Background] Pioro-Boisset M, Esdaile JM, Fitzcharles MA. Alternative medicine use in fibromyalgia syndrome. Arthritis Care Res. 1996 Feb;9(1):13-7. doi: 10.1002/art.1790090105. PMID 8945108
- [Background] Richards SC, Scott DL. Prescribed exercise in people with fibromyalgia: parallel group randomised controlled trial. BMJ. 2002 Jul 27;325(7357):185. doi: 10.1136/bmj.325.7357.185. PMID 12142304
- [Background] Russell IJ, Kamin M, Bennett RM, Schnitzer TJ, Green JA, Katz WA. Efficacy of tramadol in treatment of pain in fibromyalgia. J Clin Rheumatol. 2000 Oct;6(5):250-7. doi: 10.1097/00124743-200010000-00004. PMID 19078481
- [Background] Sayar K, Aksu G, Ak I, Tosun M. Venlafaxine treatment of fibromyalgia. Ann Pharmacother. 2003 Nov;37(11):1561-5. doi: 10.1345/aph.1D112. PMID 14565792
- [Background] Sephton SE, Salmon P, Weissbecker I, Ulmer C, Floyd A, Hoover K, Studts JL. Mindfulness meditation alleviates depressive symptoms in women with fibromyalgia: results of a randomized clinical trial. Arthritis Rheum. 2007 Feb 15;57(1):77-85. doi: 10.1002/art.22478. PMID 17266067
- [Background] Tomas-Carus P, Hakkinen A, Gusi N, Leal A, Hakkinen K, Ortega-Alonso A. Aquatic training and detraining on fitness and quality of life in fibromyalgia. Med Sci Sports Exerc. 2007 Jul;39(7):1044-50. doi: 10.1249/01.mss.0b0138059aec4. PMID 17596770
- [Background] van Koulil S, Effting M, Kraaimaat FW, van Lankveld W, van Helmond T, Cats H, van Riel PL, de Jong AJ, Haverman JF, Evers AW. Cognitive-behavioural therapies and exercise programmes for patients with fibromyalgia: state of the art and future directions. Ann Rheum Dis. 2007 May;66(5):571-81. doi: 10.1136/ard.2006.054692. Epub 2006 Aug 17. PMID 16916856
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783
- [Background] Yunus MB. Central sensitivity syndromes: a new paradigm and group nosology for fibromyalgia and overlapping conditions, and the related issue of disease versus illness. Semin Arthritis Rheum. 2008 Jun;37(6):339-52. doi: 10.1016/j.semarthrit.2007.09.003. Epub 2008 Jan 14. PMID 18191990
- [Derived] Maindet C, Maire A, Vermorel C, Cracowski C, Rolland C, Forestier R, Comte A, Roques CF, Serra E, Bosson JL. Spa Therapy for the Treatment of Fibromyalgia: An Open, Randomized Multicenter Trial. J Pain. 2021 Aug;22(8):940-951. doi: 10.1016/j.jpain.2021.02.010. Epub 2021 Mar 4. PMID 33677113